CLINICAL TRIAL: NCT03243851
Title: Efficacy and Safety of Low Dose Temozolomide Plus Metformin as Combination Chemotherapy Compared With Low Dose Temozolomide Plus Placebo in Patient With Recurrent or Refractory Glioblastoma
Brief Title: Study on Low Dose Temozolomide Plus Metformin or Placebo in Patient With Recurrent or Refractory Glioblastoma
Acronym: METT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yong-Kil Hong (Other)
Collaborators: Saint Vincent's Hospital, Korea (Other); Incheon St.Mary's Hospital (Other); National Cancer Center, Korea (Other Government); Konkuk University Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Ajou University School of Medicine (Other); Severance Hospital (Other); Chonnam National University Hospital (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yong-Kil Hong, MD., PhD., Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KNOG-1501
Record Dates: First submitted 2017-07-29; First posted 2017-08-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Arm 1 : Low dose temozolomide+metformin Arm 2 : Low dose temozolomide+placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temozolomide+metformin (Experimental): Temozolomide :
  1 cycle of 4 weeks with daily dose 50mg/m2(BSA: Body Surface Area) up to 6 cycles for 24 weeks
  Metformin :
  1. 1st cycle (4 weeks)
     * 1 week(1st~7th day) = 1,000mg/day
     * 1 week(8th~14th day) = 1,500mg/day
     * 2 weeks(15th ~28th day) = 2,000mg/day
  2. 2nd to 6th cycle (20 weeks) = 2,000mg/day
  Interventions: Drug: Temozolomide+Metformin
- Temozolomide+placebo (Placebo Comparator): Temozolomide :
  1 cycle of 4 weeks with daily dose 50mg/m2(BSA: Body Surface Area) up to 6 cycles for 24 weeks
  Placebo:
  1. 1st cycle (4 weeks)
     * 1 week(1st~7th day) = 1,000mg/day
     * 1 week(8th~14th day) = 1,500mg/day
     * 2 weeks(15th~28th day) = 2,000mg/day
  2. 2nd to 6th cycle (20 weeks) = 2,000mg/day
  Interventions: Drug: Temozolomide+Placebo

INTERVENTIONS:
Drug: Temozolomide+Metformin — Low dose temozolomide+metformin for 24 weeks
  Arms: Temozolomide+metformin
Drug: Temozolomide+Placebo — Low dose temozolomide+placebo for 24 weeks
  Arms: Temozolomide+placebo

SUMMARY:
A phase 2 clinical trial for the efficacy and safety of low dose Temozolomide plus metformin as combination chemotherapy compared with low dose Temozolomide plus placebo in patient with recurrent or refractory Glioblastoma

DETAILED DESCRIPTION:
Studies will investigate the efficacy and safety of low dose Temozolomide with Metformin or placebo for the patients with recurrent or refractory Glioblastoma.

The dosage of the Metformin will follow the domestically permitted dose to minimize side effects.

The patients will be allocated randomly to arm 1(experimental) and arm 2(placebo controlled) and administered the investigational products for up to 6 cycle. Each cycle consists of 4 weeks.

After 6 cycle(24 weeks), the patients will be checked progression and survival every 24 weeks up to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Progressive or recurrent Glioblastoma conformed by histopathological or radiological diagnosis. Progressive or recurrent Glioblastoma during or after standard therapy (Temozolomide after Temozolomide and radiation therapy; Stupp regimen) after histopathological diagnosis of Glioblastoma Recurrence or progression is diagnosed according to histopathological diagnosis or revised RANO(Response Assessment in Neuro-Oncology) criteria c
2. Karnofsky performance status(KPS) ≥ 60%
3. Age ≥ 19 years old
4. At least 4 weeks after operation or chemotherapy
5. Normal in hematological finding, liver and kidney function

   * Hematology ANC > 1.500/mm³, Platelet > 100,000/mm³, WBC > 3×10^9/L, Hemoglobin > 9g/dL
   * Liver function Total Bilirubin level ≤ 1.5×ULN(in case of isolated hyperbilirubinemia ≤2.5 x ULN) AST / ALT < 2.5×ULN
   * Renal function Serum creatinine ≤ 1.5mg/dL
6. Be informed of the nature of the study and obtained a written informed consent
7. A legal representative agrees to the trial when a subject is unable to communicate smoothly due to neurologic defect
8. If a fertile woman who has been confirmed negative to a urine or blood pregnancy test within 28 days prior to the trial

Exclusion Criteria:

1. Pregnant or breast feeding
2. Cancer history within 5 years excluding cancer in the skin cells and cervix
3. Active infections within two weeks
4. Leptomeningeal metastasis
5. Patients diagnosed with diabetes
6. Hypersensitive or intolerance to Metformin
7. Patients who are currently taking Metformin, sulfonylureas, thiazolidinediones, and insulin, regardless of reason
8. Other serious diseases or medical conditions that include :

   * Patients who suffer from unstable heart disease despite treatment.
   * Patients having a heart attack within 6 months prior to the start of trial
   * Patients who suffer from severe nerve or psychosis that includes dementia or strokes.
   * Patients with an uncontrolled infection
   * Patient with uncontrolled hypertension, congestive heart failure, unstable angina, or incomplete arrhythmia
9. Those who have participated in other clinical trials may not recover from the toxicity of the treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of progression-free survival obtained from progression-free survival curve | 24 weeks
  Comparison of progression-free survival obtained from progression-free survival curve

SECONDARY OUTCOMES:
Response Rate | 4 weeks, 8 weeks, 16 weeks, 24 weeks thereafter every 24 weeks up to 96 weeks
  Tumor Response Rate
Tumor control probability | 4 weeks, 8 weeks, 16 weeks, 24 weeks thereafter every 24 weeks up to 96 weeks
  Tumor control probability
6 month progression free survival | 24 weeks
  6 month progression free survival
6 month overall survival | 24 weeks
  6 month overall survival
Assessment of the quality of life of cancer patients | 4 weeks, 8 weeks, 16 weeks, 24 weeks
  EORTC QLQ-C30 and EORTC QLQ-BN20

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Kil Hong, MD.,PhD., Principal Investigator — Seoul St. Mary's Hospital
Locations (12):
- South Korea (12):
  - National Cancer Center Korea, Ilsan, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Incheon St. Mary's Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Saint Vincent's Hospital, Korea, Suwon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoon WS, Chang JH, Kim JH, Kim YJ, Jung TY, Yoo H, Kim SH, Ko YC, Nam DH, Kim TM, Kim SH, Park SH, Lee YS, Yim HW, Hong YK, Yang SH. Efficacy and safety of metformin plus low-dose temozolomide in patients with recurrent or refractory glioblastoma: a randomized, prospective, multicenter, double-blind, controlled, phase 2 trial (KNOG-1501 study). Discov Oncol. 2023 Jun 6;14(1):90. doi: 10.1007/s12672-023-00678-3. PMID 37278858